CLINICAL TRIAL: NCT06091696
Title: The Effect of Inspiratory Muscle Training on Respiratory Muscle Strength, Functional Capacity, Fatigue, and Stress in Breast Cancer Patients Undergoing Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Inspiratory Muscle Training on Breast Cancer Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoniem Ibrahim, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2023-367
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Post-operative Breast Cancer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: a parallel model with 2 groups of study and control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Concealed allocation will be performed by a researcher who will not be involved in the treatment of assessment. Permuted blocks will be used to ensure an equal 1:1 allocation ratio. Due to the nature of the study, the assessor and the data analyzer will be blindfolded (double-blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Inspiratory muscle training will be conducted using a pressure threshold loading device (Threshold Inspiratory Muscle Training, Respironics, Pittsburg, PA, USA). Using a spring-loaded one-way valve, this device provides air flow-independent resistance to inspiration at a detectable intensity. Patients will start training with a maximum inspiratory pressure (MIP) of 40%. The training intensity will be adjusted every week based on the MIP measurement.
  Interventions: Other: inspiratory muscle training; Other: Aerobic exercises
- control group (Active Comparator): 5 minutes of warming up and a similar time for cooling down in addition to light aerobic activity will be performed by the patients in both groups. Aerobic exercise training will be done through selected activities for 30 minutes /3 times per week for 8 weeks.
  Interventions: Other: Aerobic exercises

INTERVENTIONS:
Other: inspiratory muscle training — inspiratory muscle training will be done by using a pressure threshold loading device (Threshold Inspiratory Muscle Training, Respironics, Pittsburg, PA, USA). By using a spring-loaded one-way valve, this device provides air flow-independent resistance to inspiration at a detectable intensity.
  Arms: study group
Other: Aerobic exercises — Exercise training sessions under the supervision of an experienced physiotherapist were conducted for 30 minutes, 3 times per week, with intensity ranging between 13 and 15 on the rated perceived exertion scale (RPE).
  Other Names: exercises

SUMMARY:
This study will address the female patients who are exposed to surgery after breast cancer. strength training for the inspiratory muscles will be applied in addition to the traditional care including physical therapy that will be compared to the effect of the traditional care alone on multiple outcome measures such as muscle strength, function, fatigue, and stress.

DETAILED DESCRIPTION:
Saudi Arabia reported 24,485 new cases of cancer in 2018 with 10518 cancer deaths. There were genetic, hormonal, lifestyle, obesity, and environmental risk factors associated with different cancer types.

Many of the side effects of cancer and its treatments are burdensome and significantly impact the quality-of-life quality. Exercise before, during, and after cancer treatment provides numerous beneficial outcomes such as improving physical capacity, muscle power, and psychological status. Exercise is a valuable therapeutic tool for lowering acute, long-term, and late adverse effects of cancer.

For breast cancer patients, physiotherapy is a crucial component of treatment. The physical therapy exercise program helps patients regain fitness, reduce pain, and reduce side effects caused by different cancer treatment methods. Respiratory physiotherapy is a useful procedure for maintaining and improving functional capacity, quality of life, and post-treatment sequelae after breast cancer management, which is a combination of strategies aimed at preventing, treating, and stabilizing cardiorespiratory disorders in adults.

This study aimed to evaluate the effectiveness of inspiratory muscle training in post-surgical breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative breast cancer female patients
* Age ≥40 years
* All patients with Eastern Cooperative Oncology Group performance status score ≤ 2
* Having to undergo primary treatment with surgery

Exclusion Criteria:

* Severe anemia (Hb ≤ 8 g/dL)
* Presence of underlying chronic cardiac or respiratory disease
* severe infection, neurologic or muscular diseases prohibiting physical activity
* uncontrolled and/or extensive brain metastases, or bone metastases that were assessed to pose a risk of pathological fractures from exercising
* Contraindications descriped by the physician

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with a past history of breast cancer who underwent surgical treatment
Enrollment: 47 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength by Maximal inspiratory pressure MIP | at baseline
  Measurement of MIP will be performed using a portable electronic respiratory mouth pressure meter device (Micro RPM, Micro Medical Ltd, Kent, UK), which is a reliable and valid tool for the measurement of MIP. The MIP will be measured by deep inspiration through the mouthpiece only from the residual volume after maximal expiration. Leaning forward will not allowed during testing as it can overestimate the measurement values
Inspiratory muscle strength by Maximal inspiratory pressure MIP | after the end of the treatment (after 8 weeks)
  Measurement of MIP will be performed using a portable electronic respiratory mouth pressure meter device (Micro RPM, Micro Medical Ltd, Kent, UK), which is a reliable and valid tool for the measurement of MIP. The MIP will be measured by deep inspiration through the mouthpiece only from the residual volume after maximal expiration. Leaning forward will not allowed during testing as it can overestimate the measurement values
Inspiratory muscle strength by Maximal inspiratory pressure MIP | at follow up (3 months after the end of the treatment)
  Measurement of MIP will be performed using a portable electronic respiratory mouth pressure meter device (Micro RPM, Micro Medical Ltd, Kent, UK), which is a reliable and valid tool for the measurement of MIP. The MIP will be measured by deep inspiration through the mouthpiece only from the residual volume after maximal expiration. Leaning forward will not allowed during testing as it can overestimate the measurement values
Functional exercise capacity evaluated by a 6-minute walk test (6MWT). | baseline
  The 6-minute walk test had been clinically validated, it is used to determine the effects of therapeutic interventions and prognosis. The participants will be instructed to walk as far as possible without running in six minutes, the maximum distance covered at the end of the test will be recorded
Functional exercise capacity evaluated by a 6-minute walk test (6MWT). | after the end of the treatment (after 8 weeks)
  The 6-minute walk test had been clinically validated, it is used to determine the effects of therapeutic interventions and prognosis. The participants will be instructed to walk as far as possible without running in six minutes, the maximum distance covered at the end of the test will be recorded
Functional exercise capacity evaluated by a 6-minute walk test (6MWT). | at follow up (3 months after the end of the treatment)
  The 6-minute walk test had been clinically validated, it is used to determine the effects of therapeutic interventions and prognosis. The participants will be instructed to walk as far as possible without running in six minutes, the maximum distance covered at the end of the test will be recorded
Handgrip strength | at baseline
  Handgrip strength will be measured using handheld dynamometry. Patients have to keep the elbow of the tested side in 90 degrees of flexion and a neutral position of pronation and supination while performing the test. Both sides will be tested three times and the maximal value will be retained
Handgrip strength | after the end of the treatment (after 8 weeks)
  Handgrip strength will be measured using handheld dynamometry. Patients have to keep the elbow of the tested side in 90 degrees of flexion and a neutral position of pronation and supination while performing the test. Both sides will be tested three times and the maximal value will be retained
Handgrip strength | at follow up (3 months after the end of the treatment)
  Handgrip strength will be measured using handheld dynamometry. Patients have to keep the elbow of the tested side in 90 degrees of flexion and a neutral position of pronation and supination while performing the test. Both sides will be tested three times and the maximal value will be retained
Fatigue Assessment Scale (FAS) | baseline
  The Fatigue assessment scale (FAS) is a 10-item validated and reliable scale that will be used for evaluating symptoms of chronic fatigue.it is a self-report, paper-and-pencil measure requiring approximately 2 min for administration. Scoring each item of the FAS is answered using a five-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest
Fatigue Assessment Scale (FAS) | after the end of the treatment (after 8 weeks)
  The FAS is a 10-item validated and reliable scale that will be used for evaluating symptoms of chronic fatigue.it is a self-report, paper-and-pencil measure requiring approximately 2 min for administration. Scoring each item of the FAS is answered using a five-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest
Fatigue Assessment Scale (FAS) | at follow up (3 months after the end of the treatment)
  The FAS is a 10-item validated and reliable scale that will be used for evaluating symptoms of chronic fatigue.it is a self-report, paper-and-pencil measure requiring approximately 2 min for administration. Scoring each item of the FAS is answered using a five-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest
Perceived stress (Perceived Stress Scale pss 10) | baseline
  Is the most widely used psychological instrument for measuring the perception of stress? It is a measure of the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. Stress, Scores ranging from 0-13 would be considered low stress, and Scores ranging from 14-26 would be considered moderate stress
Perceived stress (Perceived Stress Scale pss 10) | after the end of the treatment (after 8 weeks)
  Is the most widely used psychological instrument for measuring the perception of stress? It is a measure of the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. Stress, Scores ranging from 0-13 would be considered low stress, and Scores ranging from 14-26 would be considered moderate stress
Perceived stress (Perceived Stress Scale pss 10) | at follow up (3 months after the end of the treatment)
  Is the most widely used psychological instrument for measuring the perception of stress? It is a measure of the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. Stress, Scores ranging from 0-13 would be considered low stress, and Scores ranging from 14-26 would be considered moderate stress

CONTACTS AND LOCATIONS:
Locations (1):
- Hisham Hussein, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
upon request from the funder with a reasonable need